CLINICAL TRIAL: NCT06162104
Title: Evaluation of Fatigue Severity, Mood, and Quality of Life in Post-Polio Syndrome: A Controlled Study
Brief Title: Evaluation of Fatigue Severity, Mood, and Quality of Life in Post-Polio Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH6
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Polio and Post-polio Syndrome; Fatigue; Polio
Keywords: Poliomyelitis; Fatigue; Postpoliomyelitis Syndrome
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Fatigue; Poliomyelitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-poliomyelitis syndrome group: Patients suffering from post-poliomyelitis syndrome
  Interventions: Other: No intervention
- Healthy volunteers: Control gruoup with healthy volunteers
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to investigate the differences in the severity of fatigue, impact on quality of life, and mood between individuals with post-polio syndrome and healthy volunteer groups. Additionally, the interrelationships of these parameters within the post-polio syndrome patient group will be examined. The goal is to raise awareness during the follow-up process for individuals with post-polio syndrome by questioning fatigue and mood symptoms, and to facilitate the implementation of necessary precautions.

DETAILED DESCRIPTION:
Our research is designed as a case-control study. 20 patients diagnosed with post-polio syndrome who present to the Istanbul Physical Medicine and Rehabilitation Training and Research Hospital clinics and 20 healthy volunteers will be included in the study. The sociodemographic data of patients and volunteers, such as age, gender, height, weight, body mass index, education level, and occupation, will be recorded. The age at which polio was contracted, the time elapsed since polio, and any accompanying illnesses will be documented. Additionally, if patients experience new symptoms such as pain, weakness, or fatigue, the severity of these symptoms will be assessed using the Visual Analog Scale. The frequency of falls and the presence of fractures caused by falls, ambulation method, and devices used will be noted. Muscle weakness in the extremities will be identified by applying the Manual Muscle Test through physical examination. Subsequently, the patient's current symptoms related to depression and anxiety will be evaluated using the Hospital Anxiety and Depression Scale (HADS), fatigue level will be assessed using the Fatigue Severity Scale (FSS), and quality of life will be evaluated using the Short Form-36 (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 60 with post-polio syndrome.
* Healthy volunteers aged between 18 and 60

Exclusion Criteria:

* fibromyalgia,
* chronic fatigue syndrome,
* presence of chronic decompensated cardiac, renal, and hepatic insufficiency,
* known psychiatric disorders,
* rheumatological diseases,
* presence of other known neurological diseases,
* use of medications aimed at improving physical performance or alleviating fatigue.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Individuals aged between 18 and 60 with post-polio syndrome.
  * Healthy volunteers aged between 18 and 60
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 0 day
  This scale consists of 9 items assessing the severity of fatigue and its impact on individuals. Each item is scored on a scale ranging from 0 to 7.

SECONDARY OUTCOMES:
Short Form-36 | 0 day
  This form comprises 36 items that inquire about the quality of life. Lower scores indicate a poorer condition.
Hospital Anxiety and Depression Scale | 0 day
  This scale is a 14-item assessment method, consisting of 7 questions each, designed to inquire about symptoms related to anxiety and depression in patients. As the score increases, the level of anxiety and depression worsens.
Visual Analogue Scale | 0 day
  The Visual Analog Scale is a simple measurement tool consisting of a line with endpoints representing extreme points of a characteristic, such as "No Pain" to "Worst Pain Imaginable." Respondents mark a point on the line to indicate their perception or experience of the given characteristic.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Physical Medicine and Rehabilitation Research and Training Hospital, Istanbul, Bahcelievler
  - Beylikdüzü State Hospital, Istanbul, Beylikdüzü

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gusi N, Madruga M, Gonzalez-Gonzalez MLA, Perez-Gomez J, Prieto-Prieto J. Health-related quality of life and multidimensional fitness profile in polio survivors. Disabil Rehabil. 2022 Apr;44(8):1374-1379. doi: 10.1080/09638288.2020.1804629. Epub 2020 Aug 13. PMID 32790481
- [Background] On AY, Oncu J, Atamaz F, Durmaz B. Impact of post-polio-related fatigue on quality of life. J Rehabil Med. 2006 Sep;38(5):329-32. doi: 10.1080/16501970600722395. PMID 16931464
- [Result] Bruno RL, Creange SJ, Frick NM. Parallels between post-polio fatigue and chronic fatigue syndrome: a common pathophysiology? Am J Med. 1998 Sep 28;105(3A):66S-73S. doi: 10.1016/s0002-9343(98)00161-2. PMID 9790485